CLINICAL TRIAL: NCT02625922
Title: A Multicenter, Randomized, Double-blind, Crossover Placebo-controlled Phase II Study to Assess the Effect of Serelaxin Versus Placebo on High-sensitivity Cardiac Troponin I (Hs-cTnI) Release in Patients With Chronic Heart Failure After Exercise When Used in Addition to Standard of Care
Brief Title: Study of the Effect of Serelaxin on High-sensitivity Cardiac Troponin I (Hs-cTnI) Release in Patients With Chronic Heart Failure
Acronym: RELAX-Cardio
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In view of outcome of RELAX-AHF-2 trial, the entire RLX030A project was decided to be terminated.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRLX030A2211; 2015-002673-38 (EudraCT Number)
Record Dates: First submitted 2015-12-03; First posted 2015-12-09 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-01

CONDITIONS: Chronic Heart Failure
Keywords: Serelaxin,; Chronic heart failure,; Spiroergometry,; Troponin,; New York Heart Association (NYHA) functional Class II/III,; Left ventricular ejection fraction,
MeSH Terms: interventions — serelaxin protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serelaxin followed by Placebo (Experimental): On Day 1 of treatment period 1, Serelaxin will be administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen The routine exercise assessment will commence at minute 120. In treatment period 2, on day 15 ± 1-day washout, matching placebo will be administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen.
  Interventions: Drug: Serelaxin; Drug: Placebo
- Placebo followed by Serelaxin (Experimental): On Day 1 of treatment period 1, matching placebo will be administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen The routine exercise assessment will commence at minute 120. In treatment period 2, on day 15 ± 1-day washout, Serelaxin will be administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen.
  Interventions: Drug: Serelaxin; Drug: Placebo

INTERVENTIONS:
Drug: Serelaxin — Serelaxin will be administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen
  Other Names: RLX030
Drug: Placebo — Matching placebo i.v infusion

SUMMARY:
This was a multicenter, randomized, double-blind, crossover, placebo-controlled, Phase II clinical study that evaluated the effect of serelaxin versus placebo (both in addition to SoC) on the release of hs-cTnI, in patients with CHF after an exercise testing session.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female ≥ 18 years of age, with body weight ≤ 160 Kg
* Diagnosis of stable CHF:

  * New York Heart Association (NYHA) functional Class II/III.
  * Receiving guideline-recommended treatment for CHF.
* Left ventricular ejection fraction < 45%, obtained within the last 3 months prior to screening.
* NT-proBNP > 300 ng/L in sinus rhythm or > 900 ng/L if not in sinus rhythm (determined locally).
* Ability to exercise for at least 10 to 12 minutes based on investigator's judgment.
* Systolic BP ≥ 125 mmHg at randomization
* Renal function defined as an eGFR of ≥ 25 mL/min/1.73 m^2 at screening (sMDRD formula).

Key Exclusion Criteria:

* Dyspnea primarily due to non-cardiac causes.
* Increased risk of developing hypotension during vasodilator therapy according to investigators judgement.
* Any contraindication for exercise testing and spirometry.
* Stopping of the spiroergometry at screening according to the stopping rules, unless the patient has reached maximum exercise capacity defined as carbon dioxide production/oxygen consumption (VCO2/VO2) > 1.05.
* Change in guideline-recommended CHF treatment within 1 month prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-05; Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Germany (4):
  - Novartis Investigative Site, Greifswald, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, München
- Novartis Investigative Site, Basel, Switzerland
- United Kingdom (3):
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Tyne and Wear

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were total 11 centers from 3 countries. (Germany-6, Switzerland-1, and the United Kingdom-4).
Groups:
- Serelaxin-Placebo: Subjects received serelaxin in Treatment Period 1 and placebo in Treatment Period 2.
  Serelaxin was administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen. Matching placebo was administered as an i.v infusion.
- Placebo-Serelaxin: Subjects received placebo in Treatment Period 1 and serelaxin in Treatment Period 2.
  Serelaxin was administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen. Matching placebo was administered as an i.v infusion.
Period: Overall Study
Arm/Group | Serelaxin-Placebo | Placebo-Serelaxin
Started | 14 | 12
Completed Treatment Period 1 | 12 | 10
Completed Treatment Period 2 | 11 | 8
Completed | 12 | 10
Not Completed | 2 | 2
Not completed — Non-availability of IMP | 1 | 1
Not completed — Systolic blood pressure < 125 mmHg | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Serelaxin-Placebo | Placebo-Serelaxin | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (7.62) | 66.5 (13.89) | 70.9 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 13 | 10 | 23
Weight (kg) [Mean (Standard Deviation); unit: kilogram (kg)] | 84.5 (14.19) | 83.9 (17.85) | 84.2 (15.65)
Childbearing status [Count of Participants; unit: Participants] — Number of post-menopausal participants.
  Participants | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of High Sensitivity Cardiac Troponin I (Hs-cTnI) Concentration After Exercise Compared to Placebo
Description: This cardiac biomarker measurement was obtained to determine plasma concentrations following a cardiac stress test.
Time Frame: Baseline, up to 7 hours after the start of an exercise testing session on treatment period 1 (Day 1) and treatment period 2 (Day 15+/- 1)
Population: The primary analysis of mixed model repeated measures was not performed because the validation of the primary endpoint variable hs-cTnI assay (Singulex Erenna®) was not completed because of the early termination of the study and, therefore, hs-cTnI was not analyzed.
Arm/Group | Serelaxin-Placebo | Placebo-Serelaxin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Geometric Mean of High Sensitivity Cardiac Troponin I (Hs-cTnI) Concentrations After Exercise Compared to Placebo at 4 and 5 Hours
Description: This cardiac biomarker measurement was obtained to determine plasma concentrations following a cardiac stress test.
Time Frame: 4 and 5 hours after exercise testing session
Population: The objective was not analyzed because the validation of the hs-cTnI Singulex Erenna® assay was not completed because of the early termination of the study.
Arm/Group | Serelaxin-Placebo | Placebo-Serelaxin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Log-transformed Concentration of N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) Concentrations Compared to Placebo
Description: This cardiac biomarker measurement was obtained to determine plasma concentrations following a cardiac stress test.
Time Frame: Baseline, up to 7 hours after the start of an exercise testing session on treatment period 1 (Day 1) and treatment period 2 (Day 15 +/- 1)
Population: The full analysis set (FAS) consisted of all randomized patients.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Serelaxin: Participants receiving serelaxin in Treatment Period 1 and in Treatment Period 2.
  Each participant received each of the treatments in randomized order in 2 treatment periods separated by a 15 +/- 1-day washout.
  Serelaxin was administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen.
- Placebo: Participants receiving placebo in Treatment Period 1 and in Treatment Period 2. Each participant received each of the treatments in randomized order in 2 treatment periods separated by a 15 +/- 1-day washout.
  Placebo was administered as a continuous i.v. infusion according to a weight-range adjusted dosing regimen.
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 26 | 26
pg/mL
  Baseline | 13.5026 (0.64893) | 13.6217 (0.60192)
  132 minutes | 13.5729 (0.62057) | 13.7076 (0.61612)
  180 minutes | 13.5302 (0.62107) | 13.6777 (0.61118)
  240 minutes | 13.5673 (0.68419) | 13.7011 (0.58471)
  300 minutes | 13.6103 (0.63614) | 13.7129 (0.57832)
  360 minutes | 13.6687 (0.65735) | 13.7213 (0.57366)
  420 minutes | 13.6533 (0.64776) | 13.7399 (0.57361)

4. Secondary Outcome: Log-transformed Concentration Values of Heart-type Fatty Acid-binding Protein (H-FABP) Concentrations Compared to Placebo
Description: This cardiac biomarker measurement was obtained to determine plasma concentrations following a cardiac stress test.
Time Frame: as for outcome 3
Population: The full analysis set (FAS) consisted of all randomized patients. Patients were analyzed according to the treatment they had been assigned to at randomization.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 26 | 26
ng/mL
  Baseline | 8.8256 (0.67027) | 8.8810 (0.64372)
  132 minutes | 8.8644 (0.63646) | 8.8409 (0.67261)
  180 minutes | 8.7897 (0.62835) | 8.7955 (0.62729)
  240 minutes | 8.7718 (0.63971) | 8.8662 (0.58565)
  300 minutes | 8.7309 (0.62177) | 8.7202 (0.65890)
  360 minutes | 8.7692 (0.64920) | 8.8088 (0.59672)
  420 minutes | 8.7669 (0.65793) | 8.7329 (0.63139)

ADVERSE EVENTS:
Time Frame: Adverse Events are monitored from on or after the time of first administration of study treatment up to 30 days after the last administration were included.
Description: The safety set consisted of all patients who received any amount of study treatment and had at least one post-baseline safety assessment. 22 participants were included in the safety set because 4 randomized patients did not receive study treatment.
Groups:
- Total: Total
Arm/Group | Serelaxin | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 1/22
Other Adverse Events (participants affected / at risk) | 7/20 | 6/20 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin (N=20) | Placebo (N=20) | Total (N=22)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin (N=20) | Placebo (N=20) | Total (N=22)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 2 | 0 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early by Novartis, 19-Apr-2017. Because of the early termination of the study, the validation of the hs-cTnI assay was not completed and the primary efficacy endpoint was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e.,data from all sites)in the clinical trial.